CLINICAL TRIAL: NCT02723500
Title: A Study Evaluating Hyperpolarized 129 Xenon Magnetic Resonance Imaging in Subjects With Chronic Lung Disease
Brief Title: 129 Xenon MRI in Chronic Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROB0031
Record Dates: First submitted 2015-06-24; First posted 2016-03-30 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Lung Disease
Keywords: Magnetic Resonance Imaging; Pulmonary Function
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI at baseline and over time (Other): Patients with chronic lung disease will undergo pulmonary function tests, hyperpolarized Xenon MRI at each visit.
  Interventions: Device: Hyperpolarized Xenon MRI

INTERVENTIONS:
Device: Hyperpolarized Xenon MRI — Hyperpolarized noble gas imaging using Xenon-129 has been used to explore structural and functional relationships in the lung in patients with lung disease and healthy controls. In contrast to proton-based MRI imaging, 129Xe gas is used as a contrast agent to directly visualize the airways, and thus ventilation. Whereas the normal density of gas is too low to produce an easily detectable signal, this is overcome by artificially increasing the amount of polarization per unit volume using optical pumping.

SUMMARY:
Subjects aged 18-85 with lung disease will undergo hyperpolarized Xenon 129 (129-Xe) MRI and Pulmonary Function testing for the development of tools to evaluate the Apparent Diffusion Coefficient (ADC), ventilation defect percent (VDP) and pulmonary gas exchange measurements obtained by analysis of hyperpolarized 129-Xe MRI.

DETAILED DESCRIPTION:
Briefly, during a one to two hour visit, subjects will provide written informed consent and then undergo:

1. brief medical history and vital signs,
2. full pulmonary function tests,
3. proton MRI,
4. spin-density, diffusion weighted, and/or dissolved phase 129-Xe MRI,
5. Low-dose thoracic CT

Full pulmonary function tests including spirometry, plethysmography and diffusing capacity of carbon monoxide (DLCO), Multiple Breath Nitrogen Washout (MBNW) to measure Lung Clearance Index (LCI), and Forced Oscillation Technique (FOT) will be performed according to American Thoracic Society (ATS) guidelines. MedGraphics Elite Series, MedGraphics Corporation. St. Paul, Minnesota USA and/or nDD EasyOne Spirometer, nDD Medical Technologies Inc. Andover, Massachusetts USA will be used. All measurements will be performed in the Pulmonary Function Laboratory at Robarts Research Institute.

Subjects will be placed in the 3T Magnetic Resonance (MR) scanner with one of three 129-Xe chest coils fitted over their torso and chest. Hearing protection will be provided to each subject to muffle the noise produced by the gradient radiofrequency (RF) coils. A pulse oximeter lead will be attached to all of the subjects to monitor their heart rate and oxygen saturation. MRI will be performed for up to a period of 30 minutes. All subjects will have supplemental oxygen available via nasal cannula at a flow-rate of 2 liters per minute as a precaution in the event of oxygen desaturation. Thoracic low dose CT will be performed with the same inhalation breath-hold volume and maneuver (nitrogen gas only) used for MRI to obtain participant-specific high resolution images of lung anatomy (tissue structure and airway morphology).

ELIGIBILITY:
Inclusion Criteria:

* Subjects male and female aged 18-85 with diagnosed lung disease including but not limited to: asthma, emphysema, Chronic Obstructive Pulmonary Disease (COPD), bronchiectasis, sarcoidosis, pulmonary fibrosis, alpha 1-anti-trypsin deficiency, and lymphangioleiomyomatosis (LAM)
* Subject understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent
* Subject must be able to perform a breathhold for 16s.
* Subject is judged to be in otherwise stable health on the basis of medical history
* Subject able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have Forced Expiratory Volume at one second (FEV1) values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater.)
* FEV1 >25% predicted
* Forced Vital Capacity (FVC)> 25% predicted and >0.5 liter

Exclusion Criteria:

* Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material.
* Subject has a daytime room air oxygen saturation ≤ 92% ± 2% while supine.
* Patient is unable to perform spirometry or plethysmography maneuvers
* Subject unable to tolerate MRI due to patient size and/or known history of claustrophobia.
* Patient is pregnant or lactating
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
* Subject has an MRI incompatible device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percent (VDP) of the lung | 5 years
  VDP is a widely used noble gas MRI biomarkers that is calculated by normalizing ventilation defect volume to the thoracic cavity.

SECONDARY OUTCOMES:
Apparent Diffusion Coefficients (ADC) of the lung | 5 years
  Diffusion weighted noble gas MRI provides a way to quantify pulmonary microstructure by sensing the movements of inhaled gas atoms. The "apparent" dif fusion coefficient (ADC) during the diffusion time interval can be used to reflect the extent of alveolar restriction of gas atom movements, providing a surrogate measurement of airspace dimensions.
Dissolved phase spectroscopy measurements | 5 years
  129-Xe dissolved phase MRI data will be reconstructed using a re-gridding method. The following ratios will be determined by the area-under-the curve obtained from spectroscopy: red-blood-cell to alveolar membrane ratio (RBC:membrane); RBC to gas ratio (RBC:gas); and the membrane to gas ratio (membrane:gas). Spectroscopic signals will be used to reconstruct perfusion and alveolar membrane maps.

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada